CLINICAL TRIAL: NCT00730093
Title: The Absorption of Vitamin B12 Among Healthy Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Professor, md, Ebba Nexø, Klinisk Biokemisk Afd., Århus Universitetshospital, Århus Sygehus,
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: BH12008
Record Dates: First submitted 2008-07-11; First posted 2008-08-08 (Estimated); Last update posted 2009-08-06 (Estimated); Status verified 2009-08

CONDITIONS: Pregnancy
Keywords: Vitamin B12 absorption; Pregnancy
MeSH Terms: interventions — Vitamin B 12

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Other)
  Interventions: Dietary Supplement: B12 vitamin (Cyanocobalamin)

INTERVENTIONS:
Dietary Supplement: B12 vitamin (Cyanocobalamin) — Arm A: B12 vitamin (Cyanocobalamin)

SUMMARY:
During pregnancy the woman uses more vitamin B12, but we do not know, whether it is through increased absorption or it eats into the womans vitamin B12 deposit . Sufficient B-vitamin is crucial for the normal development af foetus during pregnancy.

In Denmark the National Board of Health recommend an intake of Folic Acid, from the day the woman wishes to be pregnant and to the 12. week of gestation, but there is no recommendation for vitamin B12. We will measure the vitamin B12 absorption with a new non-radioactive test, CobaSorb.

.

ELIGIBILITY:
Inclusion Criteria:

* the 13 week of gestation +/- 1 week (only fore pregnant women)
* Between 20- 40 years
* Northern European
* abel to read and understand danish

Exclusion Criteria:

* treatment with vitamin B12 within the last 5 years
* daily intake of vitamins that contain more than 1µg vitamin B12
* infectious disease
* systemic disease
* daily use of medicine that interferes with vitamin B12

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2008-08; Primary Completion 2009-07 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Change in vitamin B12 absorption during pregnancy, measured with CobaSorb. | 9 month

CONTACTS AND LOCATIONS:
Overall Officials: Ebba Nexø, Professor, Study Chair — Aarhus Universitetshospital, Aarhus Sygehus
Locations (1):
- Aarhus Universitetshospital, Skejby, Skejby, Jylland, Denmark